CLINICAL TRIAL: NCT07324811
Title: Effectiveness of a Home-based Cervical Motor Control Exercise Programme Versus Conventional Manual Therapy in Patients With Post-whiplash Neck Pain: a Randomised Clinical Trial.
Brief Title: Effectiveness of a Home-based Cervical Motor Control Exercise Programme Versus Conventional Manual Therapy in Patients With Post-whiplash Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia de Salamanca (Other)
Responsible Party: Principal Investigator, Jorge Velazquez, Principal Investigator, Universidad Pontificia de Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00043
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disease
Keywords: Whiplash; pain; exercise
MeSH Terms: conditions — Uterine Cervical Diseases; Whiplash Injuries; Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based cervical motor control exercise programme (Experimental): home-based cervical motor control exercise programme monitored by physiotherapists
  Interventions: Procedure: home-based cervical motor control exercise programme
- conventional physiotherapy treatment (Active Comparator): Conventional physiotherapy treatment including passive therapies (manual therapy) in the physiotherapy clinic.
  Interventions: Procedure: conventional physiotherapy treatment

INTERVENTIONS:
Procedure: home-based cervical motor control exercise programme — home-based programme of active cervical motor control exercises supervised by physiotherapists
  Arms: home-based cervical motor control exercise programme
Procedure: conventional physiotherapy treatment — Conventional physiotherapy treatment with passive therapy (manual therapy) carried out in a physiotherapy clinic.
  Arms: conventional physiotherapy treatment

SUMMARY:
Whiplash-associated disorders are a common cause of persistent neck pain following traffic accidents and are frequently associated with impairments in cervical motor control, pain, and functional disability. Therapeutic exercise aimed at restoring cervical motor control has shown promising results; however, evidence regarding the effectiveness of structured home-based exercise programs compared with conventional physiotherapy remains limited. The aim of this study was to compare the effectiveness of a home-based cervical motor control exercise program versus conventional physiotherapy in patients with whiplash-associated neck pain.

A randomized controlled trial with two parallel groups was conducted. Patients diagnosed with whiplash-associated neck pain were randomly assigned to either an experimental group performing a structured home-based cervical motor control exercise program or a control group receiving conventional physiotherapy based on manual therapy and cervical mobilization techniques. Outcome measures included pain intensity assessed using the Visual Analogue Scale, functional disability measured with the Neck Disability Index, and active cervical range of motion. Assessments were performed at baseline and after an eight-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the following criteria were included:
* Age between 18 and 65 years.
* Clinical diagnosis of post-whiplash neck pain resulting from a traffic accident.
* Symptoms lasting longer than four weeks.
* Presence of neck pain with a minimum intensity of 3 points on the Visual Analogue Scale.
* Ability to understand and follow the instructions of the home exercise programme.
* Signed informed consent.

Exclusion Criteria:

* Patients with the following conditions were excluded:
* Signs of severe neurological compromise or significant structural cervical pathology (fractures, cervical instability, myelopathy).
* History of cervical surgery.
* Rheumatic, neurological, or systemic diseases that could influence the results.
* Previous physiotherapy treatment for the same episode in the three months prior to the study.
* Pregnancy or any medical contraindication for therapeutic exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
pain | 2 months
  measured using the visual analogue pain scale (VAS) (where 0 is the least possible pain and 10 is the maximum possible pain)

SECONDARY OUTCOMES:
range of motion | 2 months
  The range of active cervical movement was assessed using goniometry, recording the movements of flexion, extension, rotation, and lateralisation of the cervical spine.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Randlov A, Ostergaard M, Manniche C, Kryger P, Jordan A, Heegaard S, Holm B. Intensive dynamic training for females with chronic neck/shoulder pain. A randomized controlled trial. Clin Rehabil. 1998 Jun;12(3):200-10. doi: 10.1191/026921598666881319. PMID 9688035
- [Result] Jordan A, Bendix T, Nielsen H, Hansen FR, Host D, Winkel A. Intensive training, physiotherapy, or manipulation for patients with chronic neck pain. A prospective, single-blinded, randomized clinical trial. Spine (Phila Pa 1976). 1998 Feb 1;23(3):311-8; discussion 319. doi: 10.1097/00007632-199802010-00005. PMID 9507618
- [Result] Bronfort G, Evans R, Nelson B, Aker PD, Goldsmith CH, Vernon H. A randomized clinical trial of exercise and spinal manipulation for patients with chronic neck pain. Spine (Phila Pa 1976). 2001 Apr 1;26(7):788-97; discussion 798-9. doi: 10.1097/00007632-200104010-00020. PMID 11295901
- [Result] Kjellman GV, Skargren EI, Oberg BE. A critical analysis of randomised clinical trials on neck pain and treatment efficacy. A review of the literature. Scand J Rehabil Med. 1999 Sep;31(3):139-52. doi: 10.1080/003655099444489. PMID 10458312